CLINICAL TRIAL: NCT05543798
Title: Vision-MR Ablation Catheter 2.0 for the Treatment of Ventricular Tachycardia
Brief Title: VT Ablation in the iCMR
Acronym: VISABL-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imricor Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISABL-VT
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Randomized (Experimental): All subjects with ventricular tachycardia associated with ischemic cardiomyopathy will undergo catheter ablation using the Vision-MR Ablation Catheter 2.0
  Interventions: Device: Vision-MR Ablation Catheter 2.0

INTERVENTIONS:
Device: Vision-MR Ablation Catheter 2.0 — Catheter ablation of ventricular tachycardia

SUMMARY:
The VISABL-VT is a prospective, single-arm, multi-center, interventional investigation of the safety and efficacy of radiofrequency (RF) ablation of ventricular tachycardia associated with ischemic cardiomyopathy performed with the Vision-MR Ablation Catheter 2.0 in the iCMR environment.

ELIGIBILITY:
Inclusion Criteria:

* Roll-in subjects only: Documentation of premature ventricular contractions indicated for ablation therapy (subjects may or may not be diagnosed with Ischemic Cardiomyopathy)
* Documented (ECG/EGM) spontaneous episode of sustained ventricular tachycardia within 6 months of the procedure
* Diagnosis of Ischemic Cardiomyopathy
* AAD therapy refractory, contraindicated, not tolerated, or not desired
* 18 years or older

Exclusion Criteria:

* Implanted with non-MR compatible medical devices or contraindicated for an MRI
* Presence of intracardiac thrombus (verified via CT/MRI/TEE/TTE within 48 hours of procedure - or at start of procedure)
* Thrombocytopenia or coagulopathy
* Mechanical mitral and/or aortic valve precluding access to the left ventricle
* Severe aortic stenosis
* Myocardial infarction requiring stent implantation within 90 days of procedure
* Previous cardiac surgery within 60 days of procedures
* Known/uncontrolled stroke risks
* Class IV Heart Failure
* Ejection Fraction (EF) < 25%
* Patients with a glomerular filtration rate (GFR) < 30
* Women who are pregnant
* Allergy to contrast agents (e.g., Gadolinium)
* Active infection
* Known or suspected myxoma
* Unstable angina
* Patients who do not tolerate anticoagulation therapy
* Previous intertribal septal patch or prosthetic atrial septal defect closure device
* Life expectancy < 12 months
* Enrollment in another study without sponsor approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | Perioperative/Periprocedural
  Absence of inducible clinical ventricular tachycardia (VT) following the last RF application with with the Vision-MR Ablation Catheter 2.0
Primary Safety Endpoint | 7 days
  Composite of any procedure or device related serious adverse events through 7 days post index ablation procedure

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint | 6 months
  Chronic success defined as 6-month freedom from recurrence of sustained VT or VT requiring intervention and freedom from new or increased dose of Class I or III antiarrhythmic drugs (AAD) at 6 months following the index ablation procedure.

CONTACTS AND LOCATIONS:
Locations (3):
- Herzzentrum Leipzig, Leipzig, Saxony, Germany
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - HagaZiekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: No